CLINICAL TRIAL: NCT00899327
Title: Molecular and Functional Characterisation of Bone Marrow Function in Normal Subjects, Myelodysplastic Syndromes (MDS) and Secondary Disorders of Heamatopoiesis
Brief Title: Biomarkers in Patients at Risk of Developing Myelodysplastic Syndrome or Other Disorders and in Healthy Participants
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Oxford University Hospitals NHS Trust (Other)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: CDR0000595855; MRC-MDS-BIO1; EU-20852
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2009-07-08 (Estimated); Status verified 2009-07

CONDITIONS: Leukemia; Myelodysplastic Syndromes
Keywords: myelodysplastic syndromes; acute myeloid leukemia
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Leukemia, Myeloid, Acute | interventions — DNA Methylation; Cytogenetic Analysis; Gene Expression Profiling; Polymerase Chain Reaction

INTERVENTIONS:
Genetic: DNA methylation analysis
Genetic: RNA analysis
Genetic: cytogenetic analysis
Genetic: gene expression analysis
Genetic: mutation analysis
Genetic: polymerase chain reaction
Genetic: protein expression analysis
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of blood and bone marrow in the laboratory from patients at risk of developing myelodysplastic syndrome may help doctors learn more about changes that occur in DNA and identify biomarkers related to disorders of the blood and bone marrow.

PURPOSE: This research study is looking at biomarkers in patients at risk of developing myelodysplastic syndrome or other disorders and in healthy participants.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To identify novel biomarkers of disease that would help in the initial diagnosis of myelodysplastic syndromes (MDS).

Secondary

* To understand the genesis of anemia in cancers.
* To identify novel biomarkers of disease that predict progression of MDS to acute myeloid leukemia.

OUTLINE: Blood and bone marrow samples are collected. Hemopoietic stem cells (HSC) and progenitor cells are isolated from samples for analysis. Some of these HSC and progenitor cells are used for functional assays. From the rest of the cells, DNA, RNA, and protein is extracted for molecular analyses, including gene mutation analysis, gene methylation assays, chromatin immunoprecipitation, microarray, and real-time polymerase chain reaction.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Must meet 1 of the following criteria:

  * Being investigated for a potential blood disorder due to abnormal blood count
  * Patients with a known blood disorder who are having a bone marrow sample taken as part of the assessment of that disorder
  * Patients undergoing hip replacement surgery at Nuffield Orthopaedic Centre, Oxford meeting the following criteria:

    * Not on treatment likely to impair bone marrow function
    * No history of having had treatment likely to have impaired bone marrow function
    * Normal blood count
  * Archived samples from patients with known blood disorder

PATIENT CHARACTERISTICS:

* See Disease Characteristics

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2007-01; Primary Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Identification of novel biomarkers of disease

SECONDARY OUTCOMES:
Identification of novel biomarkers of disease progression from myelodysplastic syndromes to acute myeloid leukemia
Comprehension of genesis of anemia in cancer

CONTACTS AND LOCATIONS:
Overall Officials: Vyas Paresh, MD, Principal Investigator — Oxford University Hospitals NHS Trust
Locations (1):
- Oxford Radcliffe Hospital, Oxford, England, United Kingdom